CLINICAL TRIAL: NCT03599349
Title: Evaluation of the Ulthera® System and Efficacy Correlation to Morphological Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-145
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2018-07

CONDITIONS: Facial and Neck Skin Laxity
MeSH Terms: conditions — Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Microfocused ultrasound w/ visualization (Experimental): Each subject to receive a full face and neck area treatment using a standard 800 line treatment with set energy levels (0.90 joules for the 4-4.5mm transducer, 0.30 joules for the 7-3.0mm/7-3.0N transducers and 0.75 joules for the 7-4.5mm transducer)
  Interventions: Device: Microfocused ultrasound w/ visualization

INTERVENTIONS:
Device: Microfocused ultrasound w/ visualization
  Other Names: Ultherapy

SUMMARY:
Evaluate if there is a correlation between efficacy results and where the Thermal Coagulation Points (TCPs) produced during a treatment with the Ulthera System make contact with anatomical layers of the skin and underlying tissues.

DETAILED DESCRIPTION:
This is a prospective, single-site, non-randomized study designed to evaluate if there is a correlation between efficacy results and where the Thermal Coagulation Points (TCPs), produced during treatment with the Ulthera System, make contact with the anatomical layers of skin and underlying tissues. The study consists of one Ultherapy treatment administered at two depths using DeepSEE transducers on the full-face and neck area. Ultrasound images will be captured at the beginning, middle and end of each treatment section during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject in good health.
2. Mild to moderate skin laxity on the area(s) to be treated.
3. Subject is pre-menopausal (treated in first week of cycle) or post-menopausal.
4. Subject forehead's sub-dermal layer is at least a depth of 4.5mm using the 7-4.5mm transducer.
5. Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
6. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
7. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if the following conditions is documented on the medical history:

   a. Bilateral tubal ligation at least six months prior to study enrollment.
8. Absence of physical or psychological conditions unacceptable to the investigator.
9. Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other NSAID prior to each study treatment and chronic use during the entire post-treatment study period. Washout period, if chronic user, for 4 weeks prior to the first treatment. After all study treatments are completed, limited acute NSAID use is allowed i.e a maximum of 2-3 doses, in any 2 weeks period.
10. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
11. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Presence of an active systemic or local skin disease that may affect wound healing.
2. Severe solar elastosis.
3. Excessive subcutaneous fat in the area(s) to be treated.
4. Excessive skin laxity on the area(s) to be treated.
5. Significant scarring in the area(s) to be treated that would interfere with assessing results.
6. Open wounds or lesions in the area(s) to be treated.
7. Severe or cystic acne on the area(s) to be treated.
8. Active implants (e.g., pacemakers or defibrillators), or metallic implants in the treatment areas (dental implants not included.)
9. Inability to understand the protocol or to give informed consent.
10. Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within four weeks prior to study participation or during the study.
11. Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
12. BMI equal to or greater than 25.
13. History of chronic drug or alcohol abuse.
14. History of autoimmune disease.
15. History of Hysterectomy.
16. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
17. Subjects who anticipate the need for inpatient surgery or overnight hospitalization during the study.
18. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
19. Concurrent enrollment in any study involving the use of investigational devices or drugs.
20. Current smoker or history of smoking in the last five years.
21. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
22. Use of long-wear makeup (lipstick, lip liner, mascara, etc.) within 48 hours of study photographs and assessments.
23. History of the following cosmetic treatments in the area(s) to be treated:

    1. Skin tightening procedure within the past year;
    2. Injectable filler of any type within the past: i. 12 months for Hyaluronic acid fillers (e.g. Restylane); ii 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse); iii. 24 months for Long-lasting Hyaluronic acid (Juvéderm Voluma) and Poly-L-Lactic acid fillers (e.g. Sculptra); iv. Ever for permanent fillers (e.g. Silicone, ArteFill)
    3. Neurotoxins within the past three months;
    4. Ablative resurfacing laser treatment;
    5. Nonablative, rejuvenative laser or light treatment within the past six months;
    6. Surgical dermabrasion or deep facial peels;
    7. Facelifts, blepharoplasty, or browlift within the past year; or
    8. Any history of contour threads.
24. History of using the following prescription medications:

    1. Accutane or other systemic retinoids within the past six months;
    2. Topical Retinoids within the past two weeks;
    3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix, dabigatran);
    4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (1):
- Clinical Testing of Beverly Hills, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Microfocused Ultrasound w/ Visualization: Subject were treated on the full-face and neck area treatment using a standard 800 line treatment with set energy levels (0.90 joules for the 4-4.5mm transducer, 0.30 joules for the 7-3.0mm/7-3.0N transducers and 0.75 joules for the 7-4.5mm transducer). Ultrasound images were captured at the beginning, middle, and end of each treatment section during treatment.
Period: Overall Study
Arm/Group | Microfocused Ultrasound w/ Visualization
Started | 20
Treated | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1
  Race: Black/African Amercican | 0
  Race: White | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Determine if There is a Correlation Between D90 Quantitative Efficacy Results of the Eyebrow and Lower Face Region With Where the TCPs Produced During Ultherapy Treatment Make Contact With Anatomical Layers of the Skin and Underlying Tissues.
Description: TCP = Thermal Coagulation Points. The average Superficial Musculo-Aponeurotic System (SMAS) depth in the eyebrow and lower face regions (cheeks, submental and submandibular) will be compared to quantitative measurement of lift in the eyebrow and submental/neck lift at day 90 post-treatment
Time Frame: Day 90 post treatment
Population: Quantitative assessment of lift was not performed due to lack of quality of pre- and post-treatment images and inconsistencies in head positioning of the subjects. A correlation analysis could therefore not be performed.
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 0

2. Secondary Outcome: Comparison of CGAIS Ratings to Average SMAS and Average Dermal Thickness of the Treated Areas to Determine if There is or is Not a Correlation.
Description: The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, will complete a CGAIS assessing overall aesthetic improvement at day 90 and 180 post-treatment. The CGAIS will be compared to average SMAS and average dermal thickness of the treated areas to determine if there is or is not a correlation.
Time Frame: Day 90 and 180 post-treatment
Population: CGAIS data was not collected. A correlation analysis could therefore not be performed.
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 0

3. Secondary Outcome: The Subject Will Complete a SGAIS Assessing Overall Aesthetic Improvement at Day 90 and 180 Post-treatment Which Will be Compared to Average SMAS and Average Dermal Thickness of the Treated Areas to Determine if There is or is Not a Correlation
Description: The subject will complete a SGAIS assessing overall aesthetic improvement at day 90 and 180 post-treatment which will be compared to average SMAS and average dermal thickness of the treated areas to determine if there is or is not a correlation.
Time Frame: Day 90 and 180 post-treatment
Population: SGAIS data was not collected. A correlation analysis could therefore not be performed.
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 0

4. Secondary Outcome: Qualitative Assessment of Overall Aesthetic Improvement Will be Compared to the Average SMAS and Average Dermal Thickness of the Treated Areas to Determine if There is or is Not a Correlation
Description: Degree of overall aesthetic improvement determined by a masked, qualitative assessment of photographs at 90 and 180 days post-treatment compared to baseline, based on level of clearance/improvement. The percent improvement will be compared to the average SMAS and average dermal thickness of the treated areas to determine if there is or is not a correlation.
  Level of improvement scale:
  1. 0 = 0% Improvement (None)
  2. 1 = < 25% Improvement (Mild)
  3. 2 = 26 to 50% Improvement (Moderate)
  4. 3 = 51 to 75% Improvement (Significant)
  5. 4 = 76 to 100% Improvement (Very Significant)
Time Frame: Day 90 and 180 post-treatment
Population: A total of 20 subjects were enrolled and treated. Of these, data on this secondary outcome was available for 20 subjects at day 90 and for 19 subjects at day 180. Correlation was analyzed for the overall duration of the study (including both D90 and D180 data).
Measure: Number; unit: Correlation coefficient
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 20
Correlation coefficient
  Dermal thickness to overall aesthetic improvement | 0.2791
  SMAS thickness to overall aesthetic improvement | -1.0156

5. Secondary Outcome: The Subject Will Complete a Patient Satisfaction Questionnaire at the 90 and 180 Day Follow-up Visits Which Will be Compared to Average SMAS and Average Dermal Thickness of the Treated Areas to Determine if There is or is Not a Correlation
Description: The subject will complete a patient satisfaction questionnaire at the 90 and 180 day follow-up visits which will be compared to average SMAS and average dermal thickness of the treated areas to determine if there is or is not a correlation.
Time Frame: Day 90 and 180 post-treatment
Population: as for outcome 4
Measure: Number; unit: Correlation coefficient
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 20
Correlation coefficient
  Dermis Depth to patient satisfaction | -2.1597
  SMAS thickness to patient satisfaction | 0.0216

6. Secondary Outcome: The Depth of Frontal Region Tissue Layers Will be Compared to the Quantitative Measurements of Lift in the Eyebrow Region to Determine if There is or is Not a Correlation.
Description: The depth of the following frontal region tissue layers; dermis, subq adipose/fibrous septae, suprafrontalis fascia, frontalis muscle and subfrontalis fascia will be compared to the quantitative measurement of lift in the eyebrow region to determine if there is or is not a correlation
Time Frame: Day 90 and 180 post-treatment
Population: Quantitative assessment of lift was not performed due to lack of consistency and usability of pre- and post-treatment images and inconsistencies in head positioning of the subjects. A correlation analysis could therefore not be performed.
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 0

7. Secondary Outcome: The Depth of the Temple Region Tissue Layers Will be Compared to the Quantitative Measurement of Lift the Eyebrow Region to Determine if There is or is Not a Correlation.
Description: The depth of the following temple region tissue layers; dermis, subq adipose/fibrous septae, SMAS and temporalis muscle will be compared to the quantitative measurements of lift in the eyebrow region to determine if there is or is not a correlation.
Time Frame: Day 90 and 180 post-treatment
Population: as for outcome 6
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 0

8. Secondary Outcome: The Depth of Cheek Tissue Layers Will be Compared to the Quantitative Measurement of Lift in the Lower Face Regions to Determine if There is or is Not a Correlation.
Description: The depth of the following cheek tissue layers; dermis, subq adipose/fibrous septae, and SMAS will be compared to the quantitative measurement of lift in the lower face regions to determine if there is or is not a correlation.
Time Frame: Day 90 and 180 post-treatment
Population: as for outcome 6
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 0

9. Secondary Outcome: The Depth of Submental Tissue Layers Will be Compared to the Quantitative Measurement of Lift in the Lower Face Regions to Determine if There is or is Not a Correlation
Description: The depth of the following submental tissue layers; dermis, subq adipose/fibrous septae, supraplatysmal fascia, platysma and subplatysmal fascia will be compared to the quantitative measurement of lift in the lower face regions to determine if there is or is not a correlation.
Time Frame: Day 90 and 180 post-treatment
Population: Quantitative assessment of lift was not performed. Lack of consistency and usability of pre- and post-treatment images and inconsistencies in head positioning of the subjects. A correlation analysis could therefore not be performed.
Arm/Group | Microfocused Ultrasound w/ Visualization
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 180 days
Arm/Group | Microfocused Ultrasound w/ Visualization
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microfocused Ultrasound w/ Visualization (N=20)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microfocused Ultrasound w/ Visualization (N=20)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Bunion operation (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No